CLINICAL TRIAL: NCT03274401
Title: Screening for Atrial Fibrillation in Pulmonary Embolism Study - SAFE-PE Study
Brief Title: Screening for Atrial Fibrillation in Pulmonary Embolism Study -SAFE-PE Study
Acronym: SAFE-PE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SAFE-PE
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation; Pulmonary Embolism
Keywords: Atrial fibrillation; Pulmonary embolism; Screening
MeSH Terms: conditions — Atrial Fibrillation; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed pulmonary embolism will be randomized to screening for atrial fibrillation or standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Arm (Active Comparator): Screening for atrial fibrillation using a hand-held ECG device (Zenicor intermittent ECG) at least twice daily for two weeks. In patients where AF is detected prolonged OAC therapy will be administered.
  Interventions: Device: Zenicor intermittent ECG device; Device: 5 day ECG patch
- Control Arm (No Intervention): Standard of care

INTERVENTIONS:
Device: Zenicor intermittent ECG device — At least two weeks of screening twice daily for atrial fibrillation using intermittent ECG recordings, and prolonged use of OAC-therapy if atrial fibrillation is detected
  Other Names: Oral anticoagulant therapy prolonged (if AF detected)
  Arms: Screening Arm
Device: 5 day ECG patch — Selection of device for monitoring clinicians' choice
  Other Names: Oral anticoagulant therapy prolonged if AF detected
  Arms: Screening Arm

SUMMARY:
Patients with newly diagnosed pulmonary embolism and high thromboembolic risk will be randomized to screening for atrial fibrillation or standard of care using intermittent ECG registration for at least two weeks.

DETAILED DESCRIPTION:
Patients included in the study might be referred for an ultrasound of deep vein thrombosis unless this has already been performed. Blood will be drawn in a subset of patients to assess cardiac biomarkers, and stored in a biobank for further analysis of thrombotic biomarkers. If a computed tomography (CT) angiogram was used as diagnostic method for pulmonary embolism a radiologic review will be performed to assess presence of right atrium thrombus, with the reviewer will be blinded to the presence of atrial fibrillation (AF). In addition, an echocardiogram of the heart will be performed.

Many patients with pulmonary embolism have prolonged symptoms of dyspnoea, and palpitations. These symptoms are also described in patients with atrial fibrillation. All participants will be asked to fill out a standardized quality of life (RAND-36)-, and a symptoms questionnaire (modified European Heart Rhythm association symptom scale). Upon inclusion all patients will be reviewed for factors predisposing to PE such as recent surgery, or illness requiring immobilisation within the past three months prior to index event.

After inclusion patients will be randomised to screening for atrial fibrillation or standard of care. Participants who get randomised into the screening arm will be screened for AF using a validated, handheld ECG device at least twice daily for two weeks. Participants who get AF diagnosed during the study will be referred for appropriate cardiology follow-up and the anticoagulant therapy will be changed from a fixed time to continued (subject to yearly reviews). Patients will then be followed for five years using the Swedish death registry, and the Swedish national patient registry, in combination with the national prescription registry for the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Recent pulmonary embolism (within three months)

Fulfilling Chads-Vasc criteria for life-long oral anticoagulant therapy (2 points for men, and 3 points for women), or age > 65 years

Exclusion Criteria:

* Known diagnosis of atrial fibrillation Contra-indication to oral anticoagulant therapy Provoked pulmonary embolism in sub-segmental artery only Active cancer therapy (on-going therapy, recent surgery or life-expectancy below 1 year)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 years after intervention
  Mortality in the screening arm compared to the control arm

SECONDARY OUTCOMES:
Mortality and thromboembolic events | 5 years after intervention
  Combined endpoint of mortality and thromboembolic events (stroke, transient ischemic attack, systemic embolism, deep vein thrombosis and pulmonary embolism) in the screening arm compared to the control arm

OTHER OUTCOMES:
Quality of life using RAND-36 | 1 year after inclusion
  All patients will fill in a quality of life questionnaire (RAND-36). Quality of life will be compared in patients where AF is detected compared to the group where AF is not detected in patients with PE. Quality of life will be measured using a RAND-36 questionnaire that uses questions regarding physical, mental and social wellbeing based on the World Health Organization's definition of health.
Quality of life using EHRA symptom scale | 1 year after inclusion
  Quality of life will be compared in patients where AF is detected compared to the group where AF is not detected. Quality of life will be measured using a modified European Heart Rhythm association (EHRA) symptom scale and reported as a separate outcome.
Assessment of clinical risk factors for atrial fibrillation in patients with pulmonary embolism | 1 year after inclusion
  Comparison of clinical characteristics (diagnosis of prior hypertension, diabetes mellitus type 2, vascular disease, heart failure, stroke/TIA) to identify risk factors for detection of AF in patients with PE, and use to build a risk score for AF detection. Patients in the intervention arm who had atrial fibrillation discovered after screening with intermittent ECG will be compared to participants in the intervention arm where atrial fibrillation was not discovered. Multivariable logistic regression will be used to determine which risk factors are most important in order to detect previously undetected AF in patients with pulmonary embolism.
Biomarkers as a prediction of diagnosis in pulmonary embolism | 5 years after inclusion
  The use of biomarkers to predict risk of future thromboembolic events and mortality in patients with PE. Blood will be collected from the majority of participants in the stuydy and stored in a biobank. Different biomarkers will be measured (for instance NT-proBNP, troponin, CRP and thromboembolic biomarkers) and the association between the levels of biomarkers and mortality, and thromboembolic morbitidy will be analysed using Cox proportional regression models.
The association between biomarkers and newly detected AF in patients with pulmonary embolism | 1 years after inclusion
  Biomarkers will be collected in the majority of patients. The levels of various biomarkers in the intervention group where AF was detected will be compared to participants in the intervention group where AF was not detected. Multivariable logistic regression will be used to study the association between biomarkers and the detection of AF in patients with PE.
Echocardiographic measures and their association with outcome in patients with PE | 5 years after inclusion
  Various echocardiographic parameters will be measured in all included patients. The echocardiographic measures in patients in the study who had a secondary outcome will be compared to patients who did not have a secondary outcome. Echocardiographic measures will be analysed using multivariable Cox regression analysis in order to find parameters that are associated with poor outcome.
Echocardiographic parameters and their association with newly detected AF in patients with PE | 1 years after inclusion
  In the intervention arm echocardiographic parameters will be compared for the group where AF was detected compared to the group where AF was not detected. Using multivariable logistic regression echocardiographic variables associated with the detection of atrial fibrillation in patients with pulmonary embolism will be studied.
Presence of right atrial thrombus on DT angiography in PE | 5 years after inclusion
  In participants where DT angiography was used in order to diagnose PE the images will be reviewed in order assess whether a right atrial thrombi could be detected. The outcome between participants with right atrial thrombus on DT angiography will be compared to participants who did not have right atrial thrombus on DT.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Wallén, MD PhD, Study Director — Karolinska Institutet - Danderyd Hospital; Emma Svennberg, MD PhD, Principal Investigator — Karolinska Institutet - Danderyd Hospital
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No